CLINICAL TRIAL: NCT06089915
Title: Assessing Effectiveness of Robot-assisted Upper-limb Exercise in Persons After Cervical Spinal Cord Injury
Brief Title: Effectiveness of Robot-assisted Upper-limb Exercise in Cervical SCI
Acronym: RVZU
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Rehabilitation Institute, Republic of Slovenia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: URIS202301
Record Dates: First submitted 2023-09-18; First posted 2023-10-19 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Cervical Vertebrae Injury
Keywords: spinal cord injury; upper limbs; impairment; rehabilitation
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Occupational therapy + robot-assisted exercise (Experimental): Standard occupational therapy five times per week for 90 minutes (tailored to the patient's needs and abilities) + five 30' sessions (2-3 per week) of robot-assisted exercise for fingers and hand using Amadeo device + five 30' sessions (2-3 per week) of robot-assisted exercise using Armeo Spring exoskeleton for facilitating gross movements of upper limbs
  Interventions: Behavioral: Standard occupational therapy; Device: Robot-assisted exercise using Amadeo device and Armeo Spring exoskeleton
- Occupational therapy only (Active Comparator): Standard occupational therapy five times per week for 90 minutes (tailored to the patient's needs and abilities)
  Interventions: Behavioral: Standard occupational therapy

INTERVENTIONS:
Behavioral: Standard occupational therapy — Standard occupational therapy as part of inpatient rehabilitation
Device: Robot-assisted exercise using Amadeo device and Armeo Spring exoskeleton — Exercise for fingers and hand using Amadeo device plus gross-motor exercise using Armeo Spring exoskeleton
  Arms: Occupational therapy + robot-assisted exercise

SUMMARY:
The aim of the project is to test the effectiveness of robot-assisted upper-limb exercise in persons after cervical spinal cord injury. In a randomised controlled two-arm trial, the effect of adding two types of robot-assisted upper-limb exercise to standard occupational therapy will be tested. Three primary and two secondary outcomes will be assessed using well-established measures.

DETAILED DESCRIPTION:
Unlike for persons after stroke, there is no high-quality evidence of the effectiveness of robot-assisted upper-limb exercise in persons after cervical spinal cord injury. For this reason, we are aiming to conduct a randomised trial. The trial will involve two groups of adult patients admitted to inpatient rehabilitation. One group will receive standard occupational therapy, tailored to the patient's needs and abilities, five times per week for 90 minutes. In addition to the standard occupational therapy, the other group will receive ten 30-minute session of robot-assisted exercise: five sessions of exercise for fingers and hand using a specialised device, and five sessions of gross-motor exercise using an exoskeleton. Three outcome measures will be used to comprehensively assess the patients at the beginning and at the end of the intervention, i.e., upon admission and discharge: the Graded Redefined Assessment of Strength, Sensibility and Prehension (GRASSP; general and Myelopathy version), the Spinal Cord Independence Measure (SCIM), and the Canadian Occupational Performance Measure (COPM). The progress in those measures will be compared between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* ability to move unloaded upper limbs
* at least 18 years of age
* ability to sit for one hour
* ability to understand the instructions for robot-assisted exercise

Exclusion Criteria:

* inability to sit for one hour
* presence of hospital-acquired infection that requires isolation
* bodily impairment other than spinal cord injury
* inability to understand the instructions for robot-assisted exercise

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Difference in Graded Redefined Assessment of Strength, Sensibility and Prehension Version 2 (GRASSP V2) score | Before intervention (at admission) and after the intervention (on average after 3 weeks)
  Clinical impairment measure specific to the upper limb for use after tetraplegia that measures sensorimotor and prehension function through three domains; total score for each body side ranges from 0 to 94; higher scores mean a better outcome
Difference in Graded Redefined Assessment of Strength, Sensibility and Prehension - Mielopathy (GRASSP-M) score | Before intervention (at admission) and after the intervention (on average after 3 weeks)
  Objective tool designed to characterize patients' functional impairment related to the upper limb, useful for diagnosing and quantifying mild dysfunction and monitoring patients for deterioration; total score for each body side ranges from 0 to 74; higher scores mean a better outcome

SECONDARY OUTCOMES:
Difference in Spinal Cord Independence Measure (SCIM) score | Before intervention (at admission) and after the intervention (on average after 3 weeks)
  Assessement of performance in activities of daily living and mobility for individuals with spinal cord injury; score ranges from 0 to 100; higher scores mean a better outcome
Difference in Canadian Occupational Performance Measure (COPM) results | Before intervention (at admission) and after the intervention (on average after 3 weeks)
  Individualized, client-centred outcome measure designed to capture a client's self-perception of performance in everyday living, over time; performance and satisfaction scores range from 1 to 10; higher scores mean a better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Tibor Kafel, OT, Principal Investigator — University Rehabilitation Institute, Republic of Slovenia
Locations (1):
- University Rehabilitation Institute, Republic of Slovenia, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No